CLINICAL TRIAL: NCT06388798
Title: Evaluation of the Effectiveness of Psychoeducational Training Given to Nurses Working in a Psychiatric Clinic: Randomized Controlled Study
Brief Title: Evaluation of the Effectiveness of Psychoeducational Training Given to Nurses Working in a Psychiatric Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Nermin Erdogan, PhD Nursing, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Ankara Etlik city hospital
Record Dates: First submitted 2024-02-26; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Nursing Education; Psychoeducation
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Psychoeducational training was given to the intervention group, nurses working in the Psychiatry clinic, for a total of 4 sessions, with two sessions of 50 minutes each.
  Interventions: Other: Education
- control group (No Intervention): No psychoeducational training was given

INTERVENTIONS:
Other: Education — Psychoeducational training
  Arms: intervention group

SUMMARY:
Summary:

Background One of the most important roles of psychiatric nurses, who help individuals, families and society in promoting health, preventing diseases and coping with problems, is their educational role. With its educational role, the nurse can help the patient and their family function at the best level in biopsychosocial integrity in preventing and coping with diseases through psychoeducation.

Goals This research was conducted to evaluate the effectiveness of psychoeducational training given to nurses working in a psychiatric clinic.

Design This research is a randomized controlled experimental study. Participants Participants were determined using simple randomization. The sample of the study consisted of 78 nurses (intervention = 39; control = 39) working in a psychiatric clinic in a city hospital in Turkey.

Methods Groups were determined using the simple randomization method. Psychoeducational training was given to the intervention group, nurses working in the Psychiatry clinic, for a total of 4 sessions, with two sessions of 50 minutes each. The data of the research were collected with the ;Personal Information Form; Form for evaluating the knowledge level of nurses working in the psychiatry clinic regarding psychoeducation and Perception of Adequacy Scale in Psychoeducation Program Development and Implementation. Data were analyzed using independent samples t test and two-way repeated measures analysis of variance (ANOVA).

ELIGIBILITY:
Inclusion Criteria:

* Working in a psychiatric clinic,
* Being a nurse

Exclusion Criteria:

* Not working in a psychiatric clinic

Ages: 23 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Psychoeducation program development and implementation competence perception scale. Data will be collected before and after the training program in the intervention group, and at parallel times to the intervention group in the control group. | 3 day
  The difference between the scale pretest and posttest score averages and the difference between groups over time will be examined.
Form for evaluating the knowledge level of nurses working in a psychiatric clinic regarding psychoeducation | 3 day
  The difference between pretest and posttest score averages and the change over time between groups will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Nermin Erdoğan, PHD, Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The results of the study will be published as an article in a scientific journal.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/98/NCT06388798/Prot_SAP_ICF_000.pdf